CLINICAL TRIAL: NCT05563441
Title: Safety and Effectiveness of Laparoscopic Colorectal Resection in Elderly Patients With Colorectal Cancer
Brief Title: Laparoscopic Colorectal Resection in Elderly
Status: Completed | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Director of Gastrointestinal Surgery department, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: OAMBP-03
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
Keywords: laparoscopy; laparotomy; elderly
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic surgery: Patients over 70 years old underwent laparoscopic colorectal resection were enrolled.
  Interventions: Procedure: laparoscopic surgery
- laparotomic surgery: Patients over 70 years old underwent laparotomic colorectal resection were enrolled.

INTERVENTIONS:
Procedure: laparoscopic surgery — Patients over 70 years old underwent laparoscopic or laparotomic colorectal resection were enrolled.
  Groups: laparoscopic surgery

SUMMARY:
This is a nested cohort study of OAMBP-01. Patients over 70 years old were enrolled into the data-analysis.

The purpose of this study was to examine the feasibility and safety of laparoscopic colorectal resection in elderly patients from a single center, and to explore if there are advantages in laparoscopic surgery.

DETAILED DESCRIPTION:
Surgical resection remains the primary treatment for CRC. Despite advancements in surgical techniques, treating elderly cancer patients remains challenging for surgeons. Perioperative risk increases as elderly patients are susceptible to cardiovascular and respiratory diseases. In addition, it has been demonstrated that elderly individuals come with more locally advanced tumor and are more likely to have obstructive or disseminated disease at the time of presentation. In addition, aging diminishes a person's physiological capacity to withstand a major operation. Therefore, surgeons preferred to choose laparotomic colorectal resection to reduce surgical duration and morbidity..

The benefits of laparoscopic colorectal resections over laparotomic surgery have been clearly demonstrated in the general population. However, previous clinical trials comparing surgical approach between laparoscopy and laparotomy restricted the patient's age <75 years, we have limited information on short- and long-term safety and efficacy of elderly patients underwent laparoscopic colorectal resection.

The purpose of this study was to examine the feasibility and safety of laparoscopic colorectal resection in elderly patients from a single center, and to explore if there are advantages in laparoscopic surgery.

This is a nested cohort study of OAMBP-01. Patients over 70 years old were enrolled into the data-analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient underwent elective laparoscopic or laparotomic colorectal resection for cancer treatment; 2. Patient baseline characteristics and surgical information were available; 3. Patients with complete follow-up data.

Exclusion Criteria:

* 1. Emergency surgery for causes including bowel obstruction, bleeding, or perforation; 2. Multiple primary malignancies; 3. Failure to follow-up.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This is a nested cohort study of OAMBP-01, patients over 70 years old underwent laparotomic surgery were enrolled into the data analysis, compared with the laparotomic colorectal resection in the same time period. All eligible patients were identified by searching the database of the Gastrointestinal Surgery Centre, Third Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
perioperative complications | 42 days after surgery
  include anastomotic leakage, surgical site infection, postoperative ileus, respiratory/urinary tract infection, and deep vein thrombosis (DVT)

SECONDARY OUTCOMES:
overall survival | 5 years
  long term prognosis
disease free survival | 5 years
  long term prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Purun Lei, M.D., Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun-Yat sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided